CLINICAL TRIAL: NCT04048876
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Dose-Finding Study To Evaluate The Efficacy and Safety Of CC-90001 In Subjects With Non-Alcoholic Steatohepatitis (NASH) and Liver Fibrosis
Brief Title: Study to Evaluate the Efficacy and Safety of CC-90001 in Participants With Non-alcoholic Steatohepatitis (NASH) and Liver Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-90001-NASH-001; U1111-1235-3234 (Other: WHO); 2018-004431-79 (EudraCT Number)
Record Dates: First submitted 2019-07-17; First posted 2019-08-07 (Actual); Results first posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Non-alcoholic Fatty Liver Disease; Liver Cirrhosis
Keywords: Non-Alcoholic Steatohepatitis; NASH; Non-Alcoholic Fatty Liver; Liver Fibrosis; CC-90001
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — CC-90001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CC-90001 400 mg once daily (QD) (Experimental): CC-90001 400 mg QD
  Interventions: Drug: CC-90001
- CC-90001 200 mg once daily (Experimental): CC-90001 200 mg QD
  Interventions: Drug: CC-90001
- CC-90001 100 mg once daily (Experimental): CC-90001 100 mg QD
  Interventions: Drug: CC-90001
- Placebo once daily (Placebo Comparator): Placebo QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CC-90001 — oral
  Arms: CC-90001 100 mg once daily; CC-90001 200 mg once daily; CC-90001 400 mg once daily (QD)
Drug: Placebo — oral
  Arms: Placebo once daily

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, multicenter, multinational, dose-finding study evaluating the efficacy of three treatment doses of CC-90001 compared with placebo, in Non-alcoholic Steatohepatitis (NASH) participants with Stage 2, Stage 3 liver fibrosis.

This study is designed to assess response to treatment on measures of fibrosis and other efficacy parameters. It will also assess dose response and overall safety.

ELIGIBILITY:
Inclusion Criteria:

* Key Inclusion Criteria Diagnosis of non-alcoholic steatohepatitis (NASH) with presence of Stage 2, Stage 3 fibrosis based of the non-alcoholic steatohepatitis (NASH) Clinical Research Network (CRN) Histologic Scoring System and a nonalcoholic fatty liver disease (NAFLD) Activity Score (NAS) of 4 or higher

Exclusion Criteria:

- Key Exclusion Criteria

1. History or evidence of decompensated liver disease,
2. Hepatitis and fibrosis more likely related to etiologies other than non-alcoholic steatohepatitis (NASH).
3. Participant has urine ethyl glucuronide (EtG) > 500 ng/mL at Screening.
4. History or positive screen for human immunodeficiency virus (HIV) infection or congenital or human immunodeficiency virus (HIV)-unrelated acquired immunodeficiencies (eg, common variable immunodeficiency [CVID]).
5. History of hepatitis B and/or hepatitis C.
6. History of malignancy within the last 5 years (exceptions: excised and cured basal/squamous cell skin carcinomas and cervical carcinoma in situ).
7. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (142):
- United States (64):
  - Saint Joseph's Hosptial and Medical Center - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - UC San Diego School of Medicine, La Jolla, California
  - Cedars-Sinai Comprehensive Transplant Center, Los Angeles, California
  - California Liver Research Institute, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California Davis Medical Center, Sacramento, California
  - Southern California GI & Liver Centers, San Clemente, California
  - University of Colorado, School of Medicine - Hepatology Clinic - Anschutz, Aurora, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Digestive Health Specialists, Lakewood Rch, Florida
  - Local Institution - 176, Lakewood Rch, Florida
  - University of Miami Schiff Center for Liver Diseases, Miami, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Tampa General Hospital, Tampa, Florida
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Rush University Medical Center - University Cardiovascular Surgeons, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - WestGlen Gastrointestinal Consultants, P.A., Shawnee Mission, Kansas
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - The Institute for Digestive Health & Liver Disease at Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Louis University School of Medicine, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Beth Israel Medical Center, New York, New York
  - Concorde Medical Group, New York, New York
  - New York Presbyterian Hospital - Weill-Cornell, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Local Institution - 102, Chapel Hill, North Carolina
  - UNC Hospitals GI Medicine Clinic, Chapel Hill, North Carolina
  - Duke University School of Medicine, Durham, North Carolina
  - Carolinas HealthCare System Digestive Health, Huntersville, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center - Center for Liver Diseases, Pittsburgh, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - ClinSearch LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Texas Clinical Research Institute LLC, Arlington, Texas
  - Liver Institute at Methodist Dallas, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Brooke Army Medical Center Francis Street Medical Center, Fort Sam Houston, Texas
  - Baylor College of Medicine - Baylor Heart Clinic, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Digestive Health Associates of Texas (DHAT), Rockwell, Texas
  - American Research Corporation, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Vermont Medical Center Gastro, Burlington, Vermont
  - Bon Secours Liver Institute of Hampton Roads, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - Virginia Commonwealth University School of Medicine, Richmond, Virginia
  - University of Washington Harborview Medical Center, Seattle, Washington
  - Liver Institute Northwest PLLC, Seattle, Washington
- Australia (5):
  - University of Sydney - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - The Alfred Hospital, Melbourne, Victoria
- Canada (4):
  - University of Calgary, Cumming School of Medicine, Calgary, Alberta
  - South Edmonton Gastroenterology, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Toronto Center for Liver Disease - Francis Family Liver Clinic, Toronto, Ontario
- France (9):
  - CHU d'Angers, Angers
  - Assistance Publique - Hopitaux de Paris - Hopital Beaujon, Clichy
  - Hopital de la Croix-Rousse, Lyon
  - Assistance Publique - Hopitaux de Paris - Hopital Cochin, Paris
  - Assistance Publique - Hopitaux de Paris - Hopital Universitaire Pitie Salpetriere, Paris
  - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Universitaire de Rennes - Hopital de Pontchaillou, Rennes
  - Hopital Hautepierre, Strasbourg
  - Local Institution - 356, Strasbourg
- Germany (4):
  - Universitaetsklinikum der RWTH Aachen, Aachen
  - Johann Wolfgang Goethe University Hospital, Frankfurt am Main
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Universitaetsklinikum Muenster, Münster
- Japan (26):
  - Hamamatsu University Hospital, Hamamatsu
  - Local Institution - 604, Hamamatsu
  - Local Institution - 608, Kashihara
  - Nara Medical University Hospital, Kashihara
  - Local Institution - 601, Kawasaki
  - Shin-Yurigaoka General Hospital, Kawasaki
  - Kurume University Hospital, Kurume, Fukuoka
  - Local Institution - 607, Kurume, Fukuoka
  - Local Institution - 615, Kyoto
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Japanese Red Cross Musashino Hospital, Musashino
  - Local Institution - 602, Musashino
  - Aichi Medical University Hospital, Nagakute
  - Local Institution - 611, Nagakute
  - Local Institution - 603, Osaka-Fu
  - Osaka University Hospital OUH, Osaka-Fu
  - Local Institution - 613, Ōgaki
  - Ogaki Municipal Hospital, Ōgaki
  - Local Institution - 609, Saga
  - Saga University Hospital, Saga
  - Belland General Hospital, Sakaishi
  - Local Institution - 605, Sakaishi
  - Local Institution - 612, Suita
  - Saiseikai Suita Hospital, Suita
  - Local Institution - 600, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
- Poland (8):
  - Katowice (DRS)Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Samodzielny Publiczny Centralny Szpital Kliniczny Im Prof. Kornela Gibinskiego, Katowice
  - Krakow Medical Center LLC, Krakow
  - Lodz (DRS)Synexus Polska Sp. Z o.o. Oddzial w Lodzi, Lodz
  - Wojewodzki Specjalistyczny Szpital im. dr Wladyslawa Bieganskiego, Lodz
  - ID Clinic, Mysłowice
  - Local Institution - 453, Mysłowice
  - Synexus SCM Sp. z o.o. Oddz. Warszawa, Warsaw
- South Korea (7):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Hanyang University Seoul Hospital, Seoul
  - Korea University Hospital at Guro, Seoul
  - Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (5):
  - Hospital Val d'Hebron, Barcelona
  - University Hospital of Girona Dr. Josep Trueta, Girona
  - Parc Tauli Hospital Universitari, Sabadell (Barcelona)
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Virgen del Rocio, Seville
- United Kingdom (10):
  - University of Birmingham Institute of Biomedical Research, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrooke's Hospital, Cambridge
  - Local Institution - 558, Hardwick
  - North Tees (DRS) Synexus North Teesside Clinical Research Centre, Hardwick
  - Local Institution - 556, Hexham
  - Synexus Hexham Clinical Research Centre, Hexham (DRS), Hexham
  - Kings College Hospital, London
  - Chelsea and Westminster Hospital NHS Foundation Trust - Chelsea and Westminster Hospital (CWH), London
  - Imperial College University Trust, London
  - Local Institution - 559, London

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- CC-90001 100mg: CC-90001 100 mg PO QD
- CC-90001 200mg: CC-90001 200 mg PO QD
- CC-90001 400mg: CC-90001 400 mg PO QD
- Placebo: Placebo
Period: Placebo Controlled Phase
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Started | 13 | 15 | 13 | 15
Continuing to Follow Up | 7 | 12 | 8 | 11
Completed (= continuing to active treatment phase) | 2 | 0 | 3 | 2
Not Completed | 11 | 15 | 10 | 13
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 1
Not completed — Study Terminated by Sponsor | 10 | 12 | 10 | 12
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Active Treatment Phase
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Started | 2 | 0 | 3 | 2
Placebo to CC-90001 200mg (Participants who received placebo in the placebo-controlled phase and then received CC-90001 200mg in active treatment phase) | 0 | 0 | 0 | 1
Placebo to CC-90001 400mg (Participants who received placebo in the placebo-controlled phase and then received CC-90001 400mg in active treatment phase.) | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 3 | 2
Not completed — Study Terminated by Sponsor | 2 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo in placebo controlled phase. CC-90001 100mg, 200mg or 400mg in active treatment extension phase
- Total: Total of all reporting groups
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo | Total
Number analyzed (Participants) | 13 | 15 | 13 | 15 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (12.37) | 58.3 (9.92) | 52.1 (11.91) | 60.5 (8.20) | 56.0 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 6 | 12 | 37
  Male | 5 | 4 | 7 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 4 | 2 | 9
  Not Hispanic or Latino | 10 | 15 | 9 | 12 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 5 | 1 | 4 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 9 | 11 | 9 | 36
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve a ≥1 Stage Improvement in Liver Fibrosis Using the NASH CRN Histological Scoring System at Week 52
Description: Percentage of participants who achieve a ≥1 stage improvement in liver fibrosis using the NASH CRN Histological Scoring System at Week 52. A participant with a change of ≤ -1 from baseline in fibrosis stage is considered as an improvement responder for this endpoint.
  The NASH CRN Histologic Scoring System comprised:
  steatosis (0 to 3) lobular inflammation (0 to 3) hepatocellular ballooning (0 to 2) fibrosis disease stage (0 to 4)
  * Stage 0 - None;
  * Stage 1a - Mild (delicate) zone 3 perisinusoidal fibrosis;
  * Stage 1b - Moderate (dense) zone 3 perisinusoidal fibrosis;
  * Stage 1c - Portal/periportal fibrosis only;
  * Stage 2 - Zone 3 perisinusoidal fibrosis with portal/periportal fibrosis;
  * Stage 3 - Bridging fibrosis;
  * Stage 4 - Cirrhosis.
Time Frame: From baseline up to week 52
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 13 | 15 | 13 | 15
Percentage of Participants | 15.4 [1.92 to 45.45] | 0 [0 to 21.80] | 7.7 [0.19 to 36.03] | 6.7 [0.17 to 31.95]

2. Secondary Outcome: Percentage of Participants With no Worsening of Steatohepatitis and ≥1 Stage Improvement in Liver Fibrosis Score at Week 52
Description: Percentage of participants with no worsening of steatohepatitis and ≥1 stage improvement in liver fibrosis score at week 52 using the NASH CRN Histological Scoring System at Week 52. A participant with a change of ≥ -1 from baseline in fibrosis stage and no worsening in steatohepatitis is considered as an improvement responder for this endpoint.
  The NASH CRN Histologic Scoring System comprised:
  steatosis (0 to 3) lobular inflammation (0 to 3) hepatocellular ballooning (0 to 2) fibrosis disease stage (0 to 4)
  * Stage 0 - None;
  * Stage 1a - Mild (delicate) zone 3 perisinusoidal fibrosis;
  * Stage 1b - Moderate (dense) zone 3 perisinusoidal fibrosis;
  * Stage 1c - Portal/periportal fibrosis only;
  * Stage 2 - Zone 3 perisinusoidal fibrosis with portal/periportal fibrosis;
  * Stage 3 - Bridging fibrosis;
  * Stage 4 - Cirrhosis.
Time Frame: From baseline up to week 52
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 13 | 15 | 13 | 15
Percentage of Participants | 15.4 [1.92 to 45.45] | 0 [0 to 21.80] | 7.7 [0.19 to 36.03] | 6.7 [0.17 to 31.95]

3. Secondary Outcome: Percentage of Participants With Improvement in Total NAS
Description: Percentage of participants with an improvement of ≥ 2 points in the total NAS with improvement in more than one category of steatosis, lobular inflammation, and hepatocellular ballooning, and no worsening of liver fibrosis at Week 52. A participant with a change of ≤ -2 from baseline in total NAS, a change of ≤ -1 from baseline in more than one subscore, and a change of ≤ 0 from baseline in fibrosis stage is considered as a responder for this endpoint.
Time Frame: From baseline up to week 52
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 13 | 15 | 13 | 15
Percentage of Participants | 7.7 [0.19 to 36.03] | 6.7 [0.17 to 31.95] | 15.4 [1.92 to 45.45] | 13.3 [1.66 to 40.46]

4. Secondary Outcome: Percentage of Participants With Resolution of NASH
Description: Percentage of participants who demonstrate absence of ballooning, and lobular inflammation score of 0 or 1 at Week 52.
  Absence of ballooning is defined as a score of 0 in hepatocellular ballooning. A participant with a score of 0 in ballooning, a score of 0 or 1 in lobular inflammation is considered as a responder for this endpoint.
Time Frame: From baseline up to week 52
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 13 | 15 | 13 | 15
Percentage of Participants | 15.4 [1.92 to 45.45] | 0 [0.00 to 21.80] | 7.7 [0.19 to 36.03] | 6.7 [0.17 to 31.95]

5. Secondary Outcome: Percentage of Participants With Resolution of NASH With no Worsening of Liver Fibrosis
Description: Percentage of participants who demonstrate absence of ballooning, and lobular inflammation score of 0 or 1 and no worsening of liver fibrosis at Week 52
  Absence of ballooning is defined as a score of 0 in hepatocellular ballooning. Worsening of fibrosis stage was defined as progression of NASH CRN fibrosis stage. A participant with a score of 0 in ballooning, a score of 0 or 1 in lobular inflammation, and a change of ≤ 0 from baseline in fibrosis stage is considered as a responder for this endpoint.
Time Frame: From baseline up to week 52
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 13 | 15 | 13 | 15
Percentage of Participants | 15.4 [1.92 to 45.45] | 0 [0.00 to 21.80] | 7.7 [0.19 to 36.03] | 6.7 [0.17 to 31.95]

6. Secondary Outcome: Percentage of Participants Who Progressed to Cirrhosis
Description: Percentage of participants who progressed to cirrhosis
Time Frame: From baseline up to week 52
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 13 | 15 | 13 | 15
Percentage of Participants | 0 [0 to 24.71] | 0 [0.00 to 21.80] | 7.7 [0.19 to 36.03] | 6.7 [0.17 to 31.95]

7. Secondary Outcome: Mean Change From Baseline in Liver Biochemistry
Description: Mean change from Baseline in serum aspartate aminotransferase (AST), alanine aminotransferase (ALT) and γ-glutamyl transferase (GGT)
Time Frame: From baseline up to week 52
Population: Full Analysis Set Population at Week 52 with evaluable measures
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 2 | 0 | 3 | 2
U/L
  ALT (U/L) | 26.0 (19.80) |  | -22.3 (14.19) | -6.5 (21.92)
  AST (U/L) | 9.5 (10.61) |  | -17.0 (10.15) | 7.0 (4.24)
  GGT (U/L) | 13.0 (28.28) |  | -6.3 (5.86) | 2.5 (58.69)

8. Secondary Outcome: Mean Change From Baseline in Metabolic Parameters
Description: Mean change from baseline in total low density cholesterol (LDL) high density cholesterol (HDL), and triglycerides
Time Frame: From baseline up to week 52
Population: Full Analysis Set Population at Week 52 with evaluable measures
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 2 | 0 | 3 | 2
mmol/L
  HDL (mmol/L) | 0.005 (0.0354) |  | 0.147 (0.2155) | 0.120 (0.2687)
  LDL (mmol/L) | 0.970 (0.4525) |  | 0.623 (0.3785) | -1.395 (1.3223)
  Triglycerides (mmol/L) | -0.135 (0.0495) |  | 0.027 (0.2650) | -0.805 (0.5445)

9. Secondary Outcome: Cmax
Description: Cmax is defined as maximum plasma concentration of the drug
Time Frame: Day 1 and at Week 4
Population: PK evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 1 | 0 | 2 | 0
ng/mL
  Day 1 | 501.0 (NA) — Insufficient number of participants to calculate |  | 2938.8 (44.94) |
  Week 4: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 4 | 352.0 (NA) — Insufficient number of participants to calculate |  | 2610.0 (NA) — Insufficient number of participants to calculate |

10. Secondary Outcome: Tmax
Description: Tmax is defined is the time to maximum plasma concentration
Time Frame: Day 1 and at Week 4
Population: PK evaluable population
Measure: Median (Full Range); unit: hours
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 1 | 0 | 2 | 0
hours
  Day 1 | 2.0 [2 to 2] |  | 2.0 [2 to 2] |
  Week 4: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 4 | 2.0 [2 to 2] |  | 4.0 [4 to 4] |

11. Secondary Outcome: AUC (0-t)
Description: Area under the plasma concentration time-curve. AUC from time 0 to the last time of quantifiable concentration
Time Frame: Day 1 and at Week 4
Population: PK evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 1 | 0 | 2 | 0
h*ng/mL
  Day 1 | 2322.7 (NA) — Insufficient number of participants to calculate |  | 26803.9 (62.87) |
  Week 4: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 4 | 2530.5 (NA) — Insufficient number of participants to calculate |  | 20918.8 (NA) — Insufficient number of participants to calculate |

12. Secondary Outcome: AUC t
Description: Area under the plasma concentration time-curve. AUC over the dosing interval.
Time Frame: Day 1 and at Week 4
Population: PK evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 1 | 0 | 2 | 0
h*ng/mL
  Day 1 | 2322.7 (NA) — Insufficient number of participants to calculate |  | 27173.7 (59.71) |
  Week 4: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 4 | 2530.5 (NA) — Insufficient number of participants to calculate |  | 21182.1 (NA) — Insufficient number of participants to calculate |

13. Secondary Outcome: Apparent Total Body Clearance of the Drug
Description: Apparent total body clearance of the drug (CL/F)
Time Frame: At Week 4
Population: PK evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 1 | 0 | 2 | 0
L/h | 39.5 (NA) — Insufficient number of participants with samples to calculate geometric coefficient of variation |  | 18.9 (NA) — Insufficient number of participants with samples to calculate geometric coefficient of variation |

14. Secondary Outcome: Number of Participants With Treatment Related Safety Events
Description: Number of participants with treatment related safety events
Time Frame: From baseline up to week 52
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 13 | 15 | 13 | 15
participants
  Participants with at least one TEAE | 10 | 13 | 12 | 10
  Participants with at least one TEAE related to study drug | 4 | 5 | 10 | 3
  Participants with at least one serious TEAE | 2 | 1 | 2 | 0
  Participants with at least one serious TEAE related to study drug | 0 | 1 | 0 | 0
  Participants with at least one grade 3/4 TEAE | 2 | 1 | 2 | 1
  Participants with at least one grade 3/4 TEAE related to study drug | 0 | 1 | 0 | 0
  Participants with at least one TEAE leading to dose interruption | 2 | 1 | 2 | 0
  Participants with at least one TEAE leading to being withdrawn from study drug | 0 | 1 | 0 | 0

15. Secondary Outcome: Mean Change From Baseline of ECG Results - PR Intervals
Description: Mean change from baseline in PR interval
  PR Interval: Atrial depolarization and conduction through the AV node Normal Range: 0.12 - 0.20 (120 to 200 msec)
Time Frame: From baseline up to week 52
Population: Safety Population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 13 | 15 | 13 | 15
msec
  Week 4: number analyzed (Participants) | 11 | 13 | 10 | 12
  Week 4 | 5.8 (10.42) | -5.5 (10.18) | 3.6 (14.84) | 5.0 (19.24)
  Week 12: number analyzed (Participants) | 9 | 10 | 10 | 9
  Week 12 | 5.7 (10.32) | -2.3 (10.01) | 2.3 (21.02) | 15.2 (26.99)
  Week 24: number analyzed (Participants) | 7 | 5 | 7 | 6
  Week 24 | 4.4 (7.46) | -2.8 (3.90) | -3.7 (8.99) | 3.2 (12.75)
  Week 52: number analyzed (Participants) | 2 | 0 | 3 | 2
  Week 52 | -7.0 (9.90) |  | -7.7 (27.06) | 13.5 (10.61)

16. Secondary Outcome: Mean Change From Baseline of ECG Results - QRS Duration
Description: Mean change from baseline in QRS duration QRS Duration: Ventricular depolarization and atrial repolarization Normal Range: 0.08 to 0.10 (80 to 100 msec)
Time Frame: From baseline up to week 52
Population: Safety Population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 13 | 15 | 13 | 15
msec
  Week 4: number analyzed (Participants) | 11 | 13 | 10 | 12
  Week 4 | 0.8 (2.93) | 0.1 (5.79) | -0.1 (6.90) | -1.2 (3.59)
  Week 12: number analyzed (Participants) | 9 | 10 | 10 | 9
  Week 12 | 4.0 (3.77) | 0.7 (3.56) | -2.5 (5.38) | -2.8 (3.11)
  Week 24: number analyzed (Participants) | 7 | 5 | 7 | 6
  Week 24 | -8.7 (16.54) | 0.6 (4.77) | -2.7 (3.77) | -1.0 (3.90)
  Week 52: number analyzed (Participants) | 2 | 0 | 3 | 2
  Week 52 | -5.5 (7.78) |  | -1.3 (4.16) | 1.0 (7.07)

17. Secondary Outcome: Mean Change From Baseline of ECG Results - QT Interval
Description: Mean change from baseline in QT interval
  QT Interval: Ventricular depolarization plus ventricular repolarization Normal Range: 400 to 460 msec
Time Frame: From baseline up to week 52
Population: Safety Population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 13 | 15 | 13 | 15
msec
  Week 4: number analyzed (Participants) | 11 | 13 | 10 | 12
  Week 4 | 0.4 (19.71) | -7.6 (12.52) | -0.5 (9.47) | 1.0 (13.48)
  Week 12: number analyzed (Participants) | 9 | 10 | 10 | 9
  Week 12 | 10.6 (24.57) | -9.8 (15.48) | -2.0 (27.22) | -3.3 (17.33)
  Week 24: number analyzed (Participants) | 7 | 5 | 7 | 6
  Week 24 | 12.0 (11.55) | -11.2 (12.99) | 0.6 (22.10) | 13.5 (27.07)
  Week 52: number analyzed (Participants) | 2 | 0 | 3 | 2
  Week 52 | -6.0 (8.49) |  | -15.3 (21.73) | 8.0 (25.46)

18. Secondary Outcome: Mean Change From Baseline of ECG Results - QTcB Interval
Description: Mean change from baseline in QTcB interval
  QT Interval: Ventricular depolarization plus ventricular repolarization Normal Range: 400 to 460 msec
  QTc: QT interval corrected based on the patient's heart rate
  QTcB: An electrocardiographic finding in which the QT interval corrected for heart rate using Bazzett's formula. QTc = QT/√(RR) RR= Respiration Rate
Time Frame: From baseline up to week 52
Population: Safety Population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 13 | 15 | 13 | 15
msec
  Week 4: number analyzed (Participants) | 9 | 12 | 9 | 9
  Week 4 | -0.8 (16.18) | -2.8 (17.51) | -4.0 (15.18) | -9.3 (10.81)
  Week 12: number analyzed (Participants) | 9 | 10 | 9 | 9
  Week 12 | -0.3 (19.75) | -1.5 (10.62) | -9.6 (22.59) | 1.4 (9.25)
  Week 24: number analyzed (Participants) | 7 | 5 | 6 | 4
  Week 24 | 7.9 (10.75) | 1.2 (16.41) | 0.7 (39.65) | -11.0 (10.55)
  Week 52: number analyzed (Participants) | 2 | 0 | 3 | 2
  Week 52 | -13.0 (1.41) |  | -35.0 (9.85) | 4.5 (14.85)

19. Secondary Outcome: Mean Change From Baseline of ECG Results - QTcF Interval
Description: Mean change from baseline in QTcF interval
  QT Interval: Ventricular depolarization plus ventricular repolarization Normal Range: 400 to 460 msec
  QTc: QT interval corrected based on the patient's heart rate
  QTcF: An electrocardiographic finding in which the QT interval corrected for heart rate using Fridericia's formula. QTc = QT/∛(RR) RR = Respiration rate
Time Frame: From baseline up to week 52
Population: Safety Population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CC-90001 100mg | CC-90001 200mg | CC-90001 400mg | Placebo
Number analyzed (Participants) | 13 | 15 | 13 | 15
msec
  Week 4: number analyzed (Participants) | 8 | 13 | 10 | 12
  Week 4 | -3.9 (15.33) | -3.5 (14.45) | -1.4 (12.06) | -4.0 (10.53)
  Week 12: number analyzed (Participants) | 7 | 10 | 10 | 9
  Week 12 | 1.0 (12.33) | -4.6 (6.43) | -6.3 (21.54) | -1.4 (11.24)
  Week 24: number analyzed (Participants) | 5 | 5 | 7 | 6
  Week 24 | 9.4 (8.71) | -3.0 (10.49) | -0.9 (30.17) | 2.2 (12.67)
  Week 52: number analyzed (Participants) | 2 | 0 | 3 | 2
  Week 52 | -11.5 (3.54) |  | -27.7 (7.77) | 5.5 (0.71)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events: up to 108 weeks All-cause mortality: participants were assessed from date of randomization to study completion. All-Cause Mortality: up to 108 weeks
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- CC-90001 100 mg: CC-90001 100 mg PO QD
- CC-90001 200 mg; Active Treatment Phase CC-90001 200 mg Following Placebo: CC-90001 200 mg PO QD
- CC-90001 400 mg; Active Treatment Phase CC-90001 400 mg Following Placebo: CC-90001 400 mg PO QD
Arm/Group | CC-90001 100 mg | CC-90001 200 mg | CC-90001 400 mg | Placebo | Active Treatment Phase CC-90001 200 mg Following Placebo | Active Treatment Phase CC-90001 400 mg Following Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15 | 0/13 | 0/15 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/13 | 1/15 | 2/13 | 0/15 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 10/13 | 13/15 | 12/13 | 10/15 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC-90001 100 mg (N=13) | CC-90001 200 mg (N=15) | CC-90001 400 mg (N=13) | Placebo (N=15) | Active Treatment Phase CC-90001 200 mg Following Placebo (N=1) | Active Treatment Phase CC-90001 400 mg Following Placebo (N=1)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Spinal retrolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CC-90001 100 mg (N=13) | CC-90001 200 mg (N=15) | CC-90001 400 mg (N=13) | Placebo (N=15) | Active Treatment Phase CC-90001 200 mg Following Placebo (N=1) | Active Treatment Phase CC-90001 400 mg Following Placebo (N=1)
Allergic eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 6 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 4 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nail bed infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Occult blood positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Urine cytology abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 4 | 3 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT04048876/Prot_SAP_001.pdf